CLINICAL TRIAL: NCT06511843
Title: Examining Brief, Music Interventions for Acute Pain in the X-Ray Waiting Room
Brief Title: Music for Pain in the Waiting Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00005296
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pain Coping Information (Active Comparator): A 4-minute audio recording about common pain coping techniques (e.g., ice, rest, medication, surgery).
  Interventions: Behavioral: Pain Coping Information
- Lyrical music (Experimental): A 4-minute audio recording of Leonard Cohen's song "Hallelujah" sung by Rufus Wainwright with choral accompaniment.
  Interventions: Behavioral: Lyrical Music
- Instrumental Music (Experimental): A 4-minute audio recording of instrumental, theta wave music.
  Interventions: Behavioral: Instrumental Music

INTERVENTIONS:
Behavioral: Pain Coping Information — A 4-minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery).
  Arms: Pain Coping Information
Behavioral: Lyrical Music — A 4-minute audio recording of Leonard Cohen's song "Hallelujah" sung by Rufus Wainwright with choral accompaniment.
  Arms: Lyrical music
Behavioral: Instrumental Music — A 4-minute audio recording of instrumental, theta wave music.
  Arms: Instrumental Music

SUMMARY:
This is a single-site, three-arm, parallel-group randomized clinical trial (RCT). The clinical effects of two, 4-minute, audio-recorded, music interventions (one with lyrics and the other without) for orthopedic patients will be investigated relative to a 4-minute audio-recoding about pain psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Seeking treatment at the Tallahassee Orthopedic Center

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures.
* Other unstable illness judged by research staff to interfere with study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.
Change in Anxiety Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no anxiety and 10 representing severe anxiety,

OTHER OUTCOMES:
Change in Self-Transcendent State | Immediately before to after 4-minute audio recording
  Self-transcendent state will be measured by the three-item, state version of the validated Nondual Awareness Dimensional Assessment. These three items will be scored on a Likert scale ranging from 0-10, with higher scores representing greater self-transcendence.
Experience of Emotional Chills | Immediately after 4-minute audio recording
  Emotional chills and goosebumps will be measured with two items, each scored on a 0 to 10 Likert type scale. Higher score represent more chills/goosebumps.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided